CLINICAL TRIAL: NCT06070727
Title: Patient Satisfaction and Oral Healthy Related Quality of Life of Polyetherketoneketone and Metal Framework for Management of Maxillectomy Cases: Across Over Study
Brief Title: Polyetherketoneketone and Metal Framework for Management of Maxillectomy Cases: Across Over Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M0107023RP
Record Dates: First submitted 2023-09-20; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-07

CONDITIONS: Patient Satisfaction
Keywords: Polyetherketoneketone, Metal, Obturator
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metal framework group (Other): group A: Patients will receive metallic framework with obturator for 6 months, then the metallic obturator will be replaced by PEKK obturator for another 6 months.
  Interventions: Other: Obturator
- PEKK framework group (Other): Group B: Patients will receive PEKK obturator for 6 months, then the same patients will receive metallic framework obturator for another 6 months.
  Interventions: Other: Obturator

INTERVENTIONS:
Other: Obturator — Evaluation of patient satisfaction and oral healthy related quality of life of Polyetherketoneketone(PEKK) and metal framework for management of maxillectomy cases.

SUMMARY:
Prosthetic rehabilitation of acquired maxillary defects represents a challenging mission for both the prosthodontist and psychologically traumatized patients. These defects may be due to trauma, pathological conditions, or surgical resection of oral tumors. The resulting main problem is oronasal communication leading to impairment in mastication, swallowing, speech, and facial esthetics

DETAILED DESCRIPTION:
Maxillary obturator prostheses are usually fabricated from polymethyl methacrylate (PMMA) if the patient is completely edentulous, or from PMMA and a cast frame-work if partially edentulous. As the size of the surgical resection increases, the weight of the prosthesis also increases. Traditionally, the weight of the prosthesis has been minimized through the use of hollow bulb obturators and change of manufacturing material.

Polyetherketoneketone (PEKK) has been widely tested in a number of dental applications, such as PEKK dental implants, PEKK obturators, and PEEK RPD frameworks. PEKK has a relatively low Young's modulus of 3 to 4 GPa, which is close to that of human bones, and its tensile properties are similar to those of bone, enamel, and dentin. These properties make it a suitable material for fixed and removable prostheses.(6-8) PEKK is a lightweight material with excellent biocompatibility as it can be used in combination with Computer-aided design/computer-assisted manufacturing (CAD/CAM) in fabrication of maxillofacial prostheses.(9) So the aim of this study will be, evaluation of Patient satisfaction and oral healthy related quality of life of PEKK and metal framework for management of maxillectomy cases. The null hypothesis is that, there would be no significant difference between both frameworks.

ELIGIBILITY:
Inclusion Criteria:

The patient will be selected according to the following criteria:

* Patient with unilateral total maxillectomy.
* Patients will have sufficient number of remaining teeth.
* Free from any signs of inflammation in defect area.
* Patient 3 years after receiving radiation.
* The defect size is small or large.
* Patient with susceptibility of recurrence.

Exclusion Criteria:

* Patient is still receiving radiation.
* Defect result from trauma.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-07-04 (Estimated); Study Completion 2024-08-04 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 6 months
  Obturator functioning scale (OFS) used for evaluation of patient satisfaction, such as improvement in speech, better swallowing with the obturator, feeling and appearance of the upper lip, general feeling in the mouth, self confidence, and avoidance of social family events

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed ELSawy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No